CLINICAL TRIAL: NCT06808295
Title: Dexmedetomidine As an Effective Drug in Reducing Anesthetic Requirements in Patients Undergoing External Dacrocystorhinostomy, a Randomized Controlled Study
Brief Title: Dexmedetomidine an Effective Drug in Reducing Anesthetic Requirements in External Dacrocystorhinostomy (DCR) Patients
Acronym: DCR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Research Institute of Ophthalmology, Egypt (Other)
Responsible Party: Principal Investigator, Dina Moustafa Mohamed, Principal investigator, Research Institute of Ophthalmology, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 24-11-17-6-5
Record Dates: First submitted 2024-12-14; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Patients Undergoing External Dacrocystorhinostomy Operations; Assess Decreased Anesthetic Requirements Intraoperative
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: 2 Groups, Dexmedetomidine group and control group are assigned
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine (Active Comparator): Dexmedetomidine 0.25 microgram per kilogram is used in Dacrocystorhinostomy patients 20 minutes before induction of general anesthesia
  Interventions: Drug: Dexmedetomidine Hydrochloride
- Control (No Intervention): Fentanyl as an analgesic is used with general anesthesia in Dacrocystorhinostomy patients

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — drug will be given before induction and anesthetic doses and hemodynamics will be assessed pre- intra and postoperative
  Arms: Dexmedetomidine

SUMMARY:
Assessing the intra and postoperative hemodynamic stability in patients undergoing external dacrocystorhinostomy under general anesthesia using Dexmedetomidine as a preoperative sedation compared to traditional technique with intraoperative analgesia and assessing decreased anesthetic requirements intra and postoperative

DETAILED DESCRIPTION:
Dexmedetomidine is a highly selective alpha 2 adrenoceptor agonist, having characteristics of natural sleep like sedation, can reduce pain intensity and opioid consumption without influencing the time of recovery from general anesthesia

ELIGIBILITY:
Inclusion Criteria:

patients of both sexes 16 years to 75 years of age ASA (American society of Anesthesiologists) I-III

Exclusion Criteria:

* Pediatric age group
* ASA more than III

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Maintained hemodynamic values while reducing the anesthetic requirements | from 20 minutes after administering the drug till 2 hours after full recovery
  Measuring the heart rate and the blod pressure every 5 minutes intraoperative and for half an hour postoperative to assess hemodynamic stability

SECONDARY OUTCOMES:
Delerium | from 20 minutes after administering the drug till 2 hours after full recovery
  Reducing postoperative delirium in elderly patients

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of Ophthalmolgy, Giza, Egypt